CLINICAL TRIAL: NCT03307577
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Comparison Study to Evaluate the Safety and Efficacy of UHE-101 Cream 1% When Applied Twice Daily for 12 Weeks in Subjects With Facial Acne Vulgaris
Brief Title: A Phase 2 Safety and Efficacy Study of UHE-101 Cream in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000-8651-202
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, which means that neither the patient nor the investigator will know which cream the patient is using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UHE-101 cream, 1% (Experimental): Cream is applied twice a day
  Interventions: Drug: UHE-101 Cream
- Vehicle cream (Placebo Comparator): Cream is applied twice a day
  Interventions: Other: Vehicle Cream

INTERVENTIONS:
Drug: UHE-101 Cream — Topical cream containing investigational drug at a concentration of 1%
  Arms: UHE-101 cream, 1%
Other: Vehicle Cream — Topical cream containing no drug (i.e., placebo)
  Arms: Vehicle cream

SUMMARY:
UHE-101 cream, 1% ("UHE-101") is being developed for the topical treatment of acne vulgaris. The purpose of this study is to compare the safety and efficacy of twice daily topical application of UHE-101 cream for 12 weeks to its vehicle cream in subjects with facial acne vulgaris.

DETAILED DESCRIPTION:
The purpose of this study is to test a topical cream (UHE-101) containing 1.0% of active drug, for 12 weeks, in boys and girls, men and women, in the treatment of facial acne.

Patients who qualify for this study will apply the study cream twice daily (once in the morning and once in the evening) for 12 weeks.

Half of the patients in this study will receive UHE-101 cream and half will receive a vehicle cream that does not include an active drug (i.e., placebo). This is a double-blind study, which means that neither the patient nor the investigator will know which cream the patient is using. The study will last about 12 weeks and will involve 5 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide written informed consent/assent. A patient under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing. The parent or legal guardian must provide informed consent for the patient. If a patient becomes 18 years of age during the study, the patient must provide written informed consent at that time to continue study participation.
2. Females must be post-menopausal, surgically sterile, or use an effective method of birth control.
3. Patient has moderate to severe facial acne vulgaris.
4. Patient must be in good general health as determined by the investigator and supported by medical history, physical and Vital Signs exam.

Exclusion Criteria:

1. Females who are pregnant, lactating, or are planning to become pregnant during the study.
2. Patient has active nodulocystic acne or acne conglobate, acne fulminans, or other forms of acne (e.g., acne mechanica).
3. Patient has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
4. Patient has used any of the following topical anti-acne preparations or procedures on the face:

   * Topical anti-acne treatments including, but not limited to, over the-counter (OTC) acne cleansers or treatments, benzoyl peroxide, antibiotics, azelaic acid, dapsone, sulfa based products, corticosteroids, and salicylic acid within two weeks of Baseline;
   * Topical retinoids (e.g., tazarotene, adapalene, and tretinoin) within four weeks of Baseline;
   * Light treatments, microdermabrasion, or chemical peels within eight weeks of Baseline;
   * Other topical therapy, which may materially affect the patient's acne, in the investigator's opinion.
5. Patient has used any of the following systemic anti-acne medications:

   * Corticosteroids (including intramuscular and intralesional injections) within four weeks of Baseline. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable;
   * Antibiotics or other systemic anti-acne medications within four weeks of Baseline, with the exception of five days or less of antibiotic therapy during this period, but not within one week of Baseline;
   * Androgen receptor blockers (i.e., spironolactone or flutamide) within eight weeks of Baseline; with the exception of five days or less of spironolactone therapy during this period, but not within one week of Baseline;
   * Retinoid therapy (e.g., isotretinoin) within six months of Baseline;
   * Vitamin A supplements (greater than 10,000 units per day) within six months of Baseline;
   * Other systemic therapy, which may materially affect the patient's acne, in the investigator's opinion.
6. Patient has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the study.
7. Patient has used an investigational drug or investigational device treatment within 30 days prior to first application of the test article or is currently enrolled in an investigational drug, device, or biologic study.
8. Patient has a history of sensitivity to any of the ingredients in the test articles.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) "Success" | Week 12
  Proportion of subjects achieving success in each treatment group at Week 12 using the dichotomized IGA with success defined as a score of "clear" or "almost clear" (IGA Score of 0 or 1) and a two or more grade improvement from Baseline.
Acne Lesion Counts (Absolute Change) | Week 12
  Absolute change from Baseline in Acne Lesion Counts in each treatment group at Week 12.

SECONDARY OUTCOMES:
IGA "Success" | Week 4
  Proportion of subjects achieving success in each treatment group at Week 4.
IGA "Success" | Week 8
  Proportion of subjects achieving success in each treatment group at Week 8.
Acne Lesion Counts (Absolute Change) | Week 4
  Absolute change from Baseline in Acne Lesion Counts in each treatment group at Week 4.
Acne Lesion Counts (Absolute Change) | Week 8
  Absolute change from Baseline in Acne Lesion Counts in each treatment group at Week 8.
Acne Lesion Counts (Percent Change) | Week 4
  Percent change from Baseline in lesion counts in each treatment group at Week 4
Acne Lesion Counts (Percent Change) | Week 8
  Percent change from Baseline in lesion counts in each treatment group at Week 8
Acne Lesion Counts (Percent Change) | Week 12
  Percent change from Baseline in lesion counts in each treatment group at Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Site 02, San Diego, California, United States